CLINICAL TRIAL: NCT02062840
Title: The Brain on Whole Body Hyperthermia: A Neuroimaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Charles (Chuck) Raison, Associate Professor, Department of Psychiatry (College of Medicine) and the Norton School of Family and Consumer Sciences, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-121-670-10
Record Dates: First submitted 2014-02-07; First posted 2014-02-14 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Major Depression
Keywords: Whole Body Hyperthermia; Functional Magnetic Resonance Imaging; EEG
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Magnetic Resonance Imaging; Electrocardiography; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity whole-body infrared heating and Neuroimaging (Experimental): Subjects will have an fMRI the morning of their WBH session and and fill out study questionnaires. Following the fMRI session, the participant will undergo the WBH intervention where subjects will be induced to levels of heat that increases core body temperature to approximately 37.5-38.5 °C.temperature.
  Interventions: Device: High intensity whole-body infrared heating; Device: Functional Magnetic Resonance Imaging (fMRI) and electrocardiogram (EKG); Other: Questionnaires
- Low intensity whole-body infrared heating and (Sham Comparator): Subjects will have an fMRI the morning of their WBH session and and fill out study questionnaires. Following the fMRI session, the participant will undergo the WBH-control intervention where subjects will be induced to levels of heat that causes only a minor increase in body temperature.
  Interventions: Device: Low intensity whole-body infrared heating; Device: Functional Magnetic Resonance Imaging (fMRI) and electrocardiogram (EKG); Other: Questionnaires

INTERVENTIONS:
Device: High intensity whole-body infrared heating — The Whole Body Hyperthermia system uses water-filtered infrared-A (wIRA) heat radiation. The rise in the body's core temperature is correspondingly rapid and well-tolerated. There are two phases of the thermal challenge, 1) Irradiation phase during which the patient lies recumbent with his/her head positioned outside the tent. The wIRA irradiators are arranged above the exposed upper part of the body; and 2) Heat retention phase during which the patient lies in the chamber with the walls of the tent positioned to retain heat. Core body temperatures will be raised to those comparable to a mild fever 37.8-38.5°C.
  Arms: High intensity whole-body infrared heating and Neuroimaging
Device: Low intensity whole-body infrared heating — Attenuated heating using only heating coils at the bottom of the Heckel device. This results in only a minor increase in skin temperature and no increase in core body temperature. The participant will still feel heat and will see similar lighting and hear similar sounds as those occurring during actual WBH, and will be in the chamber for the same period of time.
  Arms: Low intensity whole-body infrared heating and
Device: Functional Magnetic Resonance Imaging (fMRI) and electrocardiogram (EKG) — A standard magnetic resonance imaging (fMRI) machine will be used to take images of the brain. An standard EKG (compatible with the fMRI machine) will be used to take measurements of cardiac vagal control.
Other: Questionnaires — Weekly questionnaires to assess changes in depression, mood, perceptions of self and quality of life will be administered.

SUMMARY:
The investigators have observed in an open trial that a single session of whole body hyperthermia (WBH) induced rapid antidepressant effects that persisted for at least a week in patients with major depression (MDD) severe enough to warrant inpatient hospitalization. In addition to reducing depression, the single session of WBH induced a prolonged reduction in mean core body temperature, consistent with basic science data from our group suggesting that hyperthermia activates a skin-to-brain pathway that have been shown in animals to be important for mood and body temperature regulation. Consistent with this known anatomy in our preliminary study in depressed patients, reductions in core body temperature were highly correlated with reductions in depressive symptoms over the same time period (one week post WBH). Moreover, patients with higher mean core body temperature prior to treatment had enhanced antidepressant effects. Because increased body temperature is an outcome of poor functioning in the skin-to-brain pathway activated by WBH our data suggests that WBH may actually sensitize this pathway in ways that promote changes in brain functioning known to promote emotional well-being. The results of our first open trial have encouraged us to conduct a larger, more rigorous placebo-controlled, double blind study of WBH for MDD, which is currently underway at the University of Arizona Medical School. Missing from our assessments in this ongoing double-blind study is any measure of the impact of WBH on brain function. The current proposal addresses ths gap in our investigative portfolio by proposing to conduct a second, randomized trial of active vs. sham WBH that will examine the impact of WBH on measures of brain function known from prior studies to be important for both depression and its treatment.

DETAILED DESCRIPTION:
The Investigators have observed in an open trial that a single session of whole body hyperthermia (WBH) induced rapid antidepressant effects that persisted for at least a week in patients with major depression (MDD) severe enough to warrant inpatient hospitalization. In addition to reducing depression, the single session of WBH induced a prolonged reduction in mean core body temperature, consistent with basic science data from our group suggesting that hyperthermia activates a skin-to-brain pathway that targets specific serotonergic nuclei in the raphe. In animal models, these nuclei have been shown to be important for mood and body temperature regultion. Consistent with this known anatomy in our preliminary study in depressed patients, reductions in core body temperature were highly correlated with reductions in depressive symptoms over the same time period (one week post WBH). Moreover, patients with higher mean core body temperature prior to treatment had enhanced antidepressant effects. Because increased body temperature is an outcome of poor functioning in the skin-to-brain pathway activated by WBH our data suggest that WBH may actually sensitize this pathway in ways that promote changes in brain functioning known to promote emotional well-being. The results of our first open trial have encouraged us to conduct a larger, more rigorous placebo-controlled, double blind study of WBH for MDD, which is currently underway at the University of Arizona Medical School. In addition to assessing effects on depressive symptoms in comparison to a sham condition, this study examines the effect of WBH on body temperature, autonomic nervous system function, thermoregulatory cooling, immune, neuroendocrine and monoamine functioning and real-world daily social behavior.

Missing from our assessments in this ongoing double-blind study is any measure of the impact of WBH on brain function. The current proposal addresses ths gap in our investigative portfolio by proposing to conduct a second, randomized trial of active vs. sham WBH that will examine the impact of WBH on measures of brain function known from prior studies to be important for both depression and its treatment. These measures will include functional magnetic resonance imaging (fMRI) analyses of resting state brain connectivity as well as assessments of concordance between subgenual anterior cingulate cortex and autonomic nervous system function assessed by electrocardiogram (EKG). Prior to these fMRI assessments a structural MRI will be obtained.

The investigators propose to conduct this fMRI/EKGtudy in 30 students (15 males/15 females) recruited from the PSYC150A1 Mass survey, which allows University of Arizona students an opportunity to serve as research subjects for course credit. These potential participants will be between the ages of 18 and 30 and will have self-reported depressive symptomatology of at least moderate severity, as reflected in a Beck Depression Inventory (BDI) II score ≥ 14. Participants will be medically healthy with no history of bipolar I disorder, schizophrenia or active substance dependence. Participants will complete questionnaires one week prior to, the day of, and one week following a single administration of either WBH or sham WBH (delivered with a 1-to-1 ratio). On the morning prior receiving WBH or sham WBH and again 24 hours later all subjects will undergo fMRI/EKG assessment. This design will allow us to evaluate the acute brain effects of WBH and to evaluate the relationship between these changes and both acute and short term (i.e. one week post treatment) improvements in mood.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-30.
* Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures.
* Fluent English Speakers (for fMRI purposes)
* Right-handed (for fMRI purposes)
* For women of child-bearing potential (i.e., one who is biologically capable of becoming pregnant), must be willing to use a medically acceptable form of birth control or practice abstinence for the duration of her participation in the trial.
* Beck Depression Inventory-II Score of ≥14 (Moderate depression)
* Normal or corrected to normal vision and normal hearing (for fMRI purposes)

Exclusion Criteria:

* Any of the following diagnoses, as identified by the intake evaluation conducted or study assessments:
* A diagnosis claustrophobia severe enough that it would impair ability to be in the Heckel HT3000 hyperthermia device and/or the fMRI machine.
* A current (or within 12 months prior to the Screening visit) diagnosis of Anorexia Nervosa or Bulimia Nervosa
* A current (within 1 month prior to screening visit) diagnosis of substance dependence
* Lifetime history of schizophrenia or bipolar I disorder
* Use of psychotropic medications within 2 weeks of screening (8 weeks for fluoxetine) except for use of benzodiazepine or non-benzodiazepine sleeping agents
* Subject has a medical condition or disorder that:
* Is unstable and clinically significant, or:
* Could interfere with the accurate assessment of safety or efficacy of treatment, including:
* individuals who are using prescription drugs that may impair thermoregulatory cooling, including diuretics, barbiturates, and beta-blockers, or antihistamines,
* individuals with cardiovascular conditions or problems (uncontrolled hypertension, congestive heart failure, or documented evidence of coronary artery disease)
* individuals with chronic conditions/diseases associated with a reduced ability initiate thermoregulatory cooling, including Parkinson's, multiple sclerosis, central nervous system tumors, and diabetes with neuropathy,
* hemophiliacs/individuals prone to bleeding,
* individuals with a fever the day of study intervention,
* individuals with hypersensitivity to heat,
* individuals with recent acute joint injury,
* individuals with enclosed infections, be they dental, in joints, or in any other tissues,
* individuals with silicone or saline implants as these can overheat and lead to burning
* Clinically significant, in the investigator's opinion, abnormal findings on screening laboratory tests or physical exam as presented to the research team.
* Need for any non-protocol psychotropic medication once enrolled, with the exception of benzodiazepine or non-benzodiazepine hypnotics used at a stable dosage.
* Women who are pregnant (HCG pregnancy test at screening, or lactating, or who plan to become pregnant during the study.
* Current participation in any clinical trial that might impact results of this one, which includes participation in another clinical trial for depression, as well as drug trials with agents that might affect mood or regulation of body temperature.
* Reasonable likelihood for non-compliance with the protocol for any other reason, in the opinion of the Investigator, prohibits enrollment of subject into the study.
* Obesity and overall size of subject. It will be up to the PI's discretion will consider BMI, waist circumference, and body fat composition when determining eligibility and safety of the individual.
* History of peripheral circulatory disease, for example peripheral vascular disease, deep vein thrombosis (DVT), or lymphedema.
* History of a cerebral vascular accident
* History of stroke, epilepsy or cerebral aneurisms
* Cancer in the last five years.
* Diabetes mellitus types I or II
* Any clinically significant autoimmune disease (compensated hypothyroidism allowed)
* Any prior history of neurological disorder, traumatic brain injury associated with an alteration of consciousness, serious medical illness that could result in cognitive impairments, and drug or alcohol dependence.
* Any potential risks for MRI, including metal fragments, implants, pins or plates, pacemakers, or metal dental work.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in acute brain effects of WBH on resting state brain connectivity and function | Change from baseline in resting state brain connectivity and one day following WBH/WBH-control Treatment.
  Functional magnetic resonance imaging (fMRI) analyses of resting state brain connectivity.
Degree of concordance of brain activity with autonomic nervous system function | Change from baseline in concordance between subgenual anteriori cingulate cortex and autonomic nervous system function and one day following WBH/WBH-control Treatment.
  Functional magnetic resonance imaging (fMRI) analyses of concordance between subgenual anterior cingulate cortex and autonomic nervous system function assessed by electrocardiogram (EKG). The investigators are specifically looking at the inter-relationship between cardiac vagal control and brain activity.

SECONDARY OUTCOMES:
Change in depression scores over time. | Seven days prior to WBH/WBH-control treatment, the day of and two days immediately following WBH/WBH-control treatment, and 7 days following WBH/WBH-control treatment.
  Percent change in scores between baseline and subsequent assessments will be assessed using the Beck Depression Inventory (BDI).
Change in Positive and Negative Affect | Seven days prior to WBH/WBH-control treatment, the day of and two days immediately following WBH/WBH-control treatment, and 7 days follwoing WBH/WBH-control treatment.
  Percent change in positive and negative affect will be assessed between baseline and subsequent assessments using the Positive and Negative Affect Schedule (PANAS)
Change in ability to function in daily life | Seven days prior to WBH/WBH-control treatment, the day of and two days immediately following WBH/WBH-control treatment, and 7 days following WBH/WBH-control treatment.
  Percent change in scores between baseline and subsequent assessments will be assessed the Sheehan Disability Scale (SDS).
Change in quality of life | Seven days prior to WBH/WBH-control treatment, the day of and two days immediately following WBH/WBH-control treatment, and 7 days following WBH/WBH-control treatment.
  Percent change in scores between baseline and subsequent assessments will be assessed using the Quality of Life and Enjoyment Scale (Q-LES).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Arizona, Department of Psychiatry, College of Medicine
Locations (1):
- University of Arizona, Tucson, Arizona, United States